CLINICAL TRIAL: NCT01672593
Title: A Randomized Controlled Trial to Evaluate Endoscopy Assisted Fibrin Glue Application in the Treatment of Low-Output ECFs
Brief Title: Glue Sealing for Patients With Low-Output ECFs
Acronym: Glue-sealing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianan Ren, Vice president of department of surgery, Jinling Hospital, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120818
Record Dates: First submitted 2012-08-19; First posted 2012-08-27 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Low-output External Gastrointestinal Fistula
Keywords: Autologous platelet rich fibrin glue;; Enterocutaneous fistulas;; Single low output GI fistulas;
MeSH Terms: conditions — Intestinal Fistula | interventions — Anti-Bacterial Agents; Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRFG treatment (Experimental): As described in our previous study, platelet-rich cryoprecipitate and thrombin were obtained from 300-400ml whole blood of each patient enrolled in the autologous PRFG(platelet-rich fibrin glue) group and then frozen at -20°C for storage. Prior to application, frozen cryoprecipitate and thrombin stored were thawed in a 37°C water bath. Aminomethylbenzoic Acid (1ml: 1mg, Sigma-Aldrich, St Louis, MO) was added into the cryoprecipitate in the volume ratio of 1:10.
  Interventions: Procedure: Endoscopy exploration and glue application; Drug: Anti-Bacterial Agents; Dietary Supplement: Nutrition support; Procedure: PRFG preparation
- Bioseal treatment (Active Comparator): The commercial fibrin sealants used in the study were purchased from Guangzhou Bioseal Biotech Co. Ltd, Guangzhou, China. Upon application, two components, fibrinogen and thrombin, were placed separately in two syringes which were joined by a Y-shaped connector. The trunk of the Y-shaped connecter was connected to a single lumen catheter.
  Interventions: Procedure: Endoscopy exploration and glue application; Drug: Anti-Bacterial Agents; Dietary Supplement: Nutrition support

INTERVENTIONS:
Procedure: Endoscopy exploration and glue application — A forward-viewing fistula-fiberscope (EndoView, Outai Medical Equipment, Shanghai, China), with 15cm length and 5mm width of fiber optical wire, was inserted into the fistula tract to accomplish endoscopic visualization. Briefly, the fistula-fiberscope assisted procedure was carried out percutaneously, allowing the exposure of internal hole and the whole tracts, followed by insertion of this catheter with distal mixing device. Upon injection, two components, fibrinogen and thrombin, were mixed together in the mixing reservoir and yield a gelatin-like glue. This procedure was repeated in patients up to 3 times within 14-day FG treatment period.
Drug: Anti-Bacterial Agents — Antibacterial therapy was given to patients with signs of systemic sepsis or local inflammation with pain.
Dietary Supplement: Nutrition support — Nutritional replacement and bowel rest via enteral or parenteral nutrition.
Procedure: PRFG preparation — As described in our previous work, platelet-rich cryoprecipitate and thrombin were obtained from 300-400ml whole blood of each patient enrolled in the PRFG group and then frozen at -20°C for storage.
  Arms: PRFG treatment

SUMMARY:
Adjuvant use of fibrin glue (FG) in the fistula tract has been shown to promote closure of low-output ECFs. The primary objectives of this study are to compare the clinical efficacy, safety of autologous platelet-rich fibrin glue (PRFG) and a commercially available fibrin sealant Bioseal® in the management of patients with low-output volume ECFs.

DETAILED DESCRIPTION:
* This is a prospective, randomized, single-centered study clinical, safety and economic outcome of ECFs patients.
* Subjects are randomized to one of 2 groups:

  * Group 1: Autologous PRFG-treatment (PRFG + SOC)
  * Group 2: Commercial FG-treatment (Bioseal® + SOC)
* Study will include three phases:

  * Phase 1: Screening, consent and enrollment
  * Phase 2: Patients will receive either PRFG, or Bioseal only for 14 days
  * Phase 3: Follow up: for patients with closed fistula within 14 days, we will follow up them for 6 months. For patients whose fistulas were still open will be treated with other therapeutic option and follow up for 6 months after closure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a single tubular ECF
* Low output volume (<200 ml/24h)
* Tract length >2cm
* Tract diameter < 1cm

Exclusion Criteria:

* Cancer-infiltrated fistula
* Abscess
* Foreign bodies
* Distal bowel obstruction
* Inflammatory bowel disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome | 14 days
  Closure time (defined as the interval between the day of enrollment and day of fistula closure), Closure rate up to 14 days, Closure rate up to 180 days, Fistula recurrence rate

SECONDARY OUTCOMES:
Safety outcome | up to 180 days
  Incidence of adverse events and severe adverse events up to 180 days (defined as an event that was fatal or life-threatening, led to additional hospitalization or disability, or required an intervention to prevent one of these outcomes)

OTHER OUTCOMES:
Economic outcome | Upon enrollment, an expected average of 1 year
  Hospital cost upon enrollment; Hospital cost during entire hospital stay; Cost between fistula onset and final outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Jinling Hospital, Nanjing, Jiangsu, China